CLINICAL TRIAL: NCT03703518
Title: Effectiveness of Mixed Reality With the Hololens System Versus Conventional Cervical Exercise Program for Asymptomatic Subjects. Crossover Pilot Study
Brief Title: Mixed Reality With Hololens® Exercise Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Hector Beltran-Alacreu, Professor, Centro Universitario La Salle
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Holo-01
Record Dates: First submitted 2018-09-18; First posted 2018-10-12 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: Mixed reality; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: cross-over pilot study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed reality (Experimental): Mixed reality exercise program using the Microsoft Hololens "Roboraid" game. This group received 6 exercise sessions over 3 weeks, 2 days/week with an interval of 48 to 72 hours between sessions, using the Microsoft Hololens "Roboraid" game. The duration of the sessions will be 10 minutes.
  Interventions: Other: Mixed reality
- Conventional exercise group (Active Comparator): Conventional exercise program in cervical region based in deep neck flexors and deep neck extensors, isometric contraction during 6-8 seconds. This group received 6 exercise sessions over 3 weeks, 2 days/week with an interval of 48 to 72 hours between sessions.
  Interventions: Other: Conventional exercise group

INTERVENTIONS:
Other: Mixed reality — This group received 6 exercise sessions over 3 weeks, 2 days/week with an interval of 48 to 72 hours between sessions, using the Microsoft Hololens "Roboraid" game. The duration of the sessions will be 10 minutes.
  Arms: Mixed reality
Other: Conventional exercise group — This group received 6 exercise sessions over 3 weeks, 2 days/week with an interval of 48 to 72 hours between sessions. This program will consist on stabilisation exercises of the cervical region, in neck deep flexors and neck deep extensors muscles to provide them with strength and resistance
  Arms: Conventional exercise group

SUMMARY:
The study design is a cross-over pilot study with 15 asymptomatic subjects. There will be 2 groups, mixed reality group and conventional cervical exercise program. Both groups received 2 sessions per week with an interval of 48 hours between them during 3 consecutive weeks.

DETAILED DESCRIPTION:
The study design is a cross-over pilot study. The study was approved by the ethical committee of the Centro Superior de Estudios Universitarios La Salle. People were recruited by referral from different places of the local community of Madrid according to the CONSORT statement (Consolidated Standards of Reporting Trials). Three assessors were trained during 300 minutes about how to perform the measurements (Investigator A) and the concerned intervention to each group (Investigator B and C). The whole procedure was conducted in the Centro Superior de Estudios Universitarios La Salle. After meeting the eligibility criteria for the study, participants were randomly allocated by an external investigator to one of the two groups:

* Mixed reality group
* Conventional Exercise group

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40,
* Not experienced any neck and upper limb symptom
* Have no significant history of chronic pain disorder,
* Did not use any medication,
* Understand, write and speak Spanish fluently.

Exclusion Criteria:

* Craniocervical pain, peripheral neuropathy or history of migraine.
* Endocrine disorders, epilepsy or any psychiatric disorder, neurological disorder.
* Surgery and a history of traumatic injuries of the upper limb

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Resistance test of the neck flexor muscles | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  To perform this test that will give us the resistance in seconds, the therapist lifts the patient's head and neck until the occipital bone is approximately 2.5 cm from the table, keeping the chin tucked into the chest.

SECONDARY OUTCOMES:
Cervical Joint Position Error Test | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  The aim of this test is to assess the subject's ability to return to the starting position after a cervical rotation movement has been performed. The patient will remain seated in a chair with a backrest. You will be given a headband with a laser pointer. At 90 cm, a stitch (a kind of target) will be placed. With the eyes closed, the participant will be asked to perform a cervical rotation and return to the starting position, as precisely as possible and without any feedback.
Evaluation of User Satisfaction with Auxiliary Device Technology (QUEST 2.0) | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  This consists of 12 questions, each one of which the participant should circle with a circle the number that best describes his or her degree of satisfaction from 1 to 5 (1 being unsatisfied and 5 very satisfied)
System Usability Scale (SUS): | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  It consists of 10 questions and the participant should dial the number that best describes their degree of satisfaction from 1 to 5 (1 being unsatisfied and 5 very satisfied)
Suitability Evaluation Questionnaire (SEQ): | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  Made up of 14 questions, one of which is an open-ended question. For the remaining questions, the participant must select the number that best fits his or her answer, from 1 to 5, range 13 to 65 points. Higher values represent more dificulty using the device. This questionnaire assesses the subject's satisfaction and also the difficulty of its use.
Q-Sense (Thermotest) | change measures (Baseline, 3 weeks, 7 weeks, 10 weeks and 14 weeks)
  Q-Sense is a validated device for the measurement of heat/cold thresholds and painful heat thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards RR, Smith MT, Stonerock G, Haythornthwaite JA. Pain-related catastrophizing in healthy women is associated with greater temporal summation of and reduced habituation to thermal pain. Clin J Pain. 2006 Oct;22(8):730-7. doi: 10.1097/01.ajp.0000210914.72794.bc. PMID 16988570
- [Background] Shahrbanian S, Ma X, Korner-Bitensky N, Simmonds MJ. Scientific evidence for the effectiveness of virtual reality for pain reduction in adults with acute or chronic pain. Stud Health Technol Inform. 2009;144:40-3. PMID 19592727
- [Background] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Background] Penasco-Martin B, de los Reyes-Guzman A, Gil-Agudo A, Bernal-Sahun A, Perez-Aguilar B, de la Pena-Gonzalez AI. [Application of virtual reality in the motor aspects of neurorehabilitation]. Rev Neurol. 2010 Oct 16;51(8):481-8. Spanish. PMID 20925030
- [Background] Beltran-Alacreu H, Lopez-de-Uralde-Villanueva I, Fernandez-Carnero J, La Touche R. Manual Therapy, Therapeutic Patient Education, and Therapeutic Exercise, an Effective Multimodal Treatment of Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2015 Oct;94(10 Suppl 1):887-97. doi: 10.1097/PHM.0000000000000293. PMID 25888653
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Background] Juul T, Langberg H, Enoch F, Sogaard K. The intra- and inter-rater reliability of five clinical muscle performance tests in patients with and without neck pain. BMC Musculoskelet Disord. 2013 Dec 3;14:339. doi: 10.1186/1471-2474-14-339. PMID 24299621
- [Background] Demers L, Monette M, Lapierre Y, Arnold DL, Wolfson C. Reliability, validity, and applicability of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) for adults with multiple sclerosis. Disabil Rehabil. 2002 Jan 10-Feb 15;24(1-3):21-30. doi: 10.1080/09638280110066352. PMID 11827151